CLINICAL TRIAL: NCT05962827
Title: Testing for Increased Lipoproteins (a) [LP(a)] in Lymphedema Patients: Li-LY
Acronym: LiLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-AOI-05; 2023-A00407-38 (Other: CHU de Nice)
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determine the prevalence of hyperlipoproteinemia (a) in a population of patients with lymphedema (Experimental): The primary endpoint will be lipoprotein (a) > 30 mg/dL, defining hyperlipoproteinemia (a).
  Interventions: Diagnostic Test: lipoprotein (a)

INTERVENTIONS:
Diagnostic Test: lipoprotein (a) — dosage of lipoprotein (a)

SUMMARY:
Lymphedema is a chronic disease that causes lymph to accumulate in the interstitial tissue. The lymphatic network is involved in the metabolism of lipids and lipoproteins, and this accumulation leads to lipid deposits in the tissues involved. The level of lipoprotein(a) [LP(a)] has been shown to be a cardiovascular risk factor, which is partly genetically determined and influenced by certain factors (chronic renal failure, statin treatment, sporting activity or a diet low in saturated fatty acids...). Plasma levels of LP(a) lipoproteins (a) are linearly associated with an increased risk of myocardial infarction and carotid and femoral vascular stenosis. We currently manage patients with primary or secondary lymphedema, whatever the etiology, in the vascular medicine and explorations unit at Nice University Hospital.

Those taking part in intensive inpatient decongestive therapy benefit from a blood test, in particular for lipids [total cholesterol, triglycerides, HDL and LDL cholesterol, apolipoproteins A and B and Lp(a)]. Our team observed an elevated Lp(a) level >30 mg/dL in 10 of the 17 patients in whom we carried out this test (whether or not dyslipidemia existed, and whether or not it was known or treated). This is a very high prevalence compared with the general population, in whom an increased level is found in 25% of patients.

In view of the impact of Lp(a) on cardiovascular risk and the involvement of the lymphatic system in lipoprotein metabolism, it seems essential to verify our preliminary results on a larger population. In this multicenter cross-sectional trial, we propose to perform Lp(a) lipoprotein assays in lymphedema patients to determine whether there is an increase in this marker in this pathological context. We will also study the concordance of this level with cardiovascular risk assessment scores such as SCORE2/SCORE2-OP and the coronary calcium score. We will look for factors influencing plasma LP(a) levels, both general factors suspected of playing a role and factors specific to lymphedema.

DETAILED DESCRIPTION:
Lymphedema is a chronic disease that causes lymph to accumulate in the interstitial tissue. The lymphatic network is involved in the metabolism of lipids and lipoproteins, and this accumulation leads to lipid deposits in the tissues involved. The level of lipoprotein(a) [LP(a)] has been shown to be a cardiovascular risk factor, which is partly genetically determined and influenced by certain factors (chronic renal failure, statin treatment, sporting activity or a diet low in saturated fatty acids...). Plasma levels of LP(a) lipoproteins (a) are linearly associated with an increased risk of myocardial infarction and carotid and femoral vascular stenosis. We currently manage patients with primary or secondary lymphedema, whatever the etiology, in the vascular medicine and explorations unit at Nice University Hospital.

Those taking part in intensive inpatient decongestive therapy benefit from a blood test, in particular for lipids [total cholesterol, triglycerides, HDL and LDL cholesterol, apolipoproteins A and B and Lp(a)]. Our team observed an elevated Lp(a) level >30 mg/dL in 10 of the 17 patients in whom we carried out this test (whether or not dyslipidemia existed, and whether or not it was known or treated). This is a very high prevalence compared with the general population, in whom an increased level is found in 25% of patients.

In view of the impact of Lp(a) on cardiovascular risk and the involvement of the lymphatic system in lipoprotein metabolism, it seems essential to verify our preliminary results on a larger population. In this multicenter cross-sectional trial, we propose to perform Lp(a) lipoprotein assays in lymphedema patients to determine whether there is an increase in this marker in this pathological context. We will also study the concordance of this level with cardiovascular risk assessment scores such as SCORE2/SCORE2-OP and the coronary calcium score. We will look for factors influencing plasma LP(a) levels, both general factors suspected of playing a role and factors specific to lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patient with primary or secondary lymphedema confirmed at consultation or in day hospital.
* Signature of informed consent.
* Person affiliated to or benefiting from a social security scheme

Exclusion Criteria:

* Person refusing informed consent.
* Pregnant or breast-feeding women (urine pregnancy test performed in women of -childbearing age).
* Patients undergoing secondary cardiovascular prevention (MI, stroke, AOMI, etc.).
* Persons deprived of their liberty by judicial or administrative decision, persons under legal protection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of hyperlipoproteinemia (a) in a population of patients with primary or secondary lymphedema | day 0
  The primary endpoint will be lipoprotein (a) > 30 mg/dL, defining hyperlipoproteinemia (a).

SECONDARY OUTCOMES:
To study the modification of the SCORE-2 /SCORE-OP index of cardiovascular risk assessment at re-evaluation, | day 5
  To study the modification of the SCORE-2 /SCORE-OP index
To study the modification of the cardiovascular risk assessment calcium score at reassessment, taking into account the presence of hyperlipoproteinemia (a). | day 5
  cardiovascular risk assessment calcium score at reassessment,

CONTACTS AND LOCATIONS:
Overall Officials: Verena FASSBENDER, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - Chu de Nice, Nice, France
  - Centre antoine lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No